CLINICAL TRIAL: NCT07048639
Title: Dosimetric Evaluation of Breathing Impact on Planning Treatment Volumne and Adjacent Organ At Risk in Breast Cancer Radiotherapy
Brief Title: Dosimetric Evaluation of Breathing Impact on PTV and Adjacent Organ At Risk in Breast Cancer Radiotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/904
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Four-Dimensional Computed Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4D-CT (Four-Dimensional Computed Tomography)
  Interventions: Diagnostic Test: 4D-CT (Four-Dimensional Computed Tomography)

INTERVENTIONS:
Diagnostic Test: 4D-CT (Four-Dimensional Computed Tomography) — To assess tumor and organ motion during breathing

SUMMARY:
The study is likely an observational study, possibly retrospective or prospective, involving patients with breast cancer undergoing radiotherapy.

DETAILED DESCRIPTION:
Patients with breast cancer scheduled for radiotherapy will be selected based on specific inclusion and exclusion criteria.

Patients will undergo imaging studies, such as computed tomography (CT) scans, to define the target volumes and OARs.

The study aims to provide insights into the dosimetric impact of breathing motion on PTV and OARs in breast cancer radiotherapy, which can inform strategies to improve treatment planning and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patient of breast cancer.
* age 25-40

Exclusion Criteria:

* Patients without breast cancer

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This research study aims to evaluate the dosimetric impact of breathing on planning treatment volume (PTV) and adjacent organs at risk (OARs) in breast cancer radiotherapy. The study seeks to quantify the effects of breathing motion on radiation dose distribution, which is crucial for ensuring effective treatment and minimizing side effects.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) Scale with scoring details | 12 Months
  The Physician's Global Assessment (PGA) scale is a tool used by physicians to evaluate the overall severity of a patient's disease. It's a subjective assessment, typically on a scale of 0 to 3 or 0 to 4, with higher scores indicating more severe disease activity. The PGA focuses on the overall disease activity, considering both the severity of active manifestations and relevant laboratory results, excluding organ damage and subjective findings unrelated to disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- INMOL hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No